CLINICAL TRIAL: NCT06347965
Title: Construction and Effect Evaluation of the Low Load Blood Flow Restriction Training Program for Lung Cancer Patients Complicated With Sarcopenia During Chemotherapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Xin Wang (Other)
Responsible Party: Sponsor-Investigator, Xin Wang, Graduate student, Zhejiang University
Organization: Zhejiang University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: IIT20220541B-R1
Record Dates: First submitted 2024-03-28; First posted 2024-04-04 (Actual); Last update posted 2024-04-04 (Actual); Status verified 2024-03

CONDITIONS: Sarcopenia; Lung Neoplasms
Keywords: lung cancer; sarcopenia; the low-load blood flow restriction training; progressive resistance training
MeSH Terms: conditions — Sarcopenia; Lung Neoplasms

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Routine care group (Control group, CON) (No Intervention): During hospitalization, patients will be given routine exercise and dietary guidance.
- Low load blood flow restriction training group (LL-BFRT) (Experimental): On the basis of routine care, participants who meet the inclusion and exclusion criteria will be guided to undergo low-load blood flow restriction training. Based on the constructed "Low load Blood Flow Restriction Training Program for Chemotherapy Stage Lung Cancer Patients with Sarcopenia", participants will be guided to undergo low-load blood flow restriction training.
  Interventions: Behavioral: Low load blood flow restriction training
- Progressive resistance training group (PRE) (Active Comparator): On the basis of routine care, progressive resistance training will be conducted on subjects who meet the inclusion and exclusion criteria, guided by the progressive resistance training program for malignant tumor patients in the "ACSM Exercise Testing and Exercise Prescription Guidelines: 10th Edition" published by the People's Health Press.
  Interventions: Behavioral: Progressive resistance training group

INTERVENTIONS:
Behavioral: Low load blood flow restriction training — Low load blood flow restriction training will be conducted on the subjects three times a week. Each training session includes upper and lower limb training, with 4 groups trained and repeated 30, 15, 15, and 15 times for each group. Train for a total of 12 weeks.The resistance strength will remain at 30% RM for weeks 1-12.
  Arms: Low load blood flow restriction training group (LL-BFRT)
Behavioral: Progressive resistance training group — The subjects will undergo progressive resistance training three days a week, three groups per day, with each group repeating 10 times. Training includes upper and lower limbs. The resistance load increases over time, with a resistance load of 30% RM for weeks 1-4, 50% RM for weeks 5-8, and 70% RM for weeks 9-12.
  Arms: Progressive resistance training group (PRE)

SUMMARY:
The goal of this clinical trial is to verify the effectiveness and safety of the low load blood flow restriction training program. The intervention effect, tolerance and compliance of low load blood flow restriction training and progressive resistance training on lung cancer patients complicated with sarcopenia during chemotherapy will be compared, in order to provide new ideas for improving or reversing sarcopenia.

The main questions it aims to answer are:

Can low load blood flow restriction training improve sarcopenia in chemotherapy induced lung cancer patients? Which training method is more effective and tolerable between low load blood flow restriction training and progressive resistance training?

Participants will be randomly divided into 3 groups：

1. Routine care group (Control group, CON): The researchers will provide participants with regular exercise and dietary guidance.
2. Low load blood flow restriction group (LL-BFRT): The researchers will provide participants with a low load blood flow restriction training program constructed by our research group.
3. Progressive resistance training group (PRE): The researchers will provide participants with progressive resistance training.

ELIGIBILITY:
Inclusion Criteria:

* The pathological diagnosis is lung cancer, and the diagnostic criteria refer to the 2023 edition of the Clinical Diagnosis and Treatment Guidelines for Lung Cancer of the Chinese Medical Association.
* Diagnosed as sarcopenia, the diagnostic criteria refer to the 2023 version of the Expert Consensus on the Diagnosis and Treatment of sarcopenia in the Elderly in China.
* Chemotherapy has been carried out and the remaining chemotherapy frequency is ≥ 4 times.
* Physical disability free, Eastern Cooperative Oncology Group Performance Status (ECOG PS) ≤ 2 points
* No language communication barriers, able to cooperate in completing scale assessments
* Expected life>6 months
* Previous irregular exercise habits
* Patients and their families have informed consent and voluntarily join
* A person who has a smartphone and can complete WeChat check-in

Exclusion Criteria:

* Merge with other malignant tumors
* There are contraindications or symptoms or diseases that affect exercise, such as uncontrolled hypertension, venous thrombosis, infection, platelet count<50 × 109/L, white blood cell count<3.0 × 109/L, hemoglobin<10 mg/dL, bleeding tendency, arrhythmia, heart failure, unstable angina, heart valve disease, chronic obstructive pulmonary disease, asthma, limb dysfunction, severe muscle, bone and joint diseases, etc
* The risk factor score table for blood flow restriction training scores>2
* During rest, blood oxygen saturation ≤ 90%
* Cannot conduct human body composition analyzer testing, such as for patients with cardiovascular stent implantation, pacemaker equipped, artificial joint replacement, or amputation
* Patients carrying PICC
* Patients with cognitive impairment and mental illness
* Patients with planned weight loss

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Actual)
Dates: Start 2023-02-01 (Actual); Primary Completion 2023-11-30 (Actual); Study Completion 2024-02-20 (Actual)

PRIMARY OUTCOMES:
Grip strength | Grip strength will be measured at 3, 6, 9, and 12 weeks after intervention
  The grip strength of the participant's preferred hand
Appendicular Skeletal Muscle Index (ASMI) | ASMI will be measured at 3, 6, 9, and 12 weeks after intervention
  Using a human body composition analyzer (ICOMEON-FI2001B) to measure the skeletal muscle mass (ASM) of the limbs, and calculating ASMI using a formula. ASMI=ASM/height^2
Step speed | Step speed will be measured at 3, 6, 9, and 12 weeks after intervention
  Measure the walking speed of 6m

SECONDARY OUTCOMES:
Body mass index (BMI) | BMI will be measured at 3, 6, 9, and 12 weeks after intervention
  Measure height and weight using height measuring instruments and scales
Quality of life for lung cancer patients | Quality of life for lung cancer patients will be measured at 3, 6, 9, and 12 weeks after intervention
  Using the QLQ-LC 43 scale to measure the quality of life in lung cancer patients
Exercise compliance | Exercise compliance will be measured at12 weeks after intervention
  This includes participation rate, interruption rate (number of missed training sessions), termination rate (termination of training before 12 weeks), and dose adjustment rate (adjustment of training load or frequency)
Exercise safety | Exercise safety will be measured at12 weeks after intervention
  Record the frequency and time of adverse events caused by exercise, such as muscle pain, joint pain, dizziness, skin bruising, etc., and calculate the incidence rate of adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Xin Wang, Principal Investigator — graduate student
Locations (1):
- The First Affiliated Hospital, Zhejiang University School of Medicine, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No